CLINICAL TRIAL: NCT05146830
Title: A Long-Term Follow-Up Study of Participants With Cystinosis Who Previously Received CTNS-RD-04
Status: Enrolling by invitation | Type: Observational
Sponsor: Stephanie Cherqui (Other)
Collaborators: California Institute for Regenerative Medicine (CIRM) (Other); Cystinosis Research Foundation (Other); Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor-Investigator, Stephanie Cherqui, Principal Investigator, University of California, San Diego
Organization: University of California, San Diego (Other)
Other Study IDs: CTNS-RD-04-LTFU01
Record Dates: First submitted 2021-10-28; First posted 2021-12-07 (Actual); Last update posted 2024-07-03 (Actual); Status verified 2024-07

CONDITIONS: Cystinosis
Keywords: Cystinosis Disease; Cell therapy; Gene therapy; Long-term follow-up
MeSH Terms: conditions — Cystinosis | interventions — Safety

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood, urine, bone marrow, and hair sample collections.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Participants with Cystinosis Disease: This is a long-term follow-up study of participants who previously received CTNS-RD-04 (single dose administration). No investigational product will be administered in this study.
  Interventions: Other: Safety and Efficacy Assessments

INTERVENTIONS:
Other: Safety and Efficacy Assessments — Safety evaluations, disease-specific assessments, and other assessments to monitor for long-term complications of gene therapy intervention.
  Other Names: Gene Therapy Intervention

SUMMARY:
This is a multinational, long-term follow-up study to assess the long-term safety and durability of CTNS-RD-04 treatment in participants who received a single dose administration of lentiviral gene therapy. No investigational product will be administered in this study. Participants will continue periodic safety and efficacy assessments in this long-term follow-up study up to 15 years from the initial date of CTNS-RD-04 infusion.

DETAILED DESCRIPTION:
Participants enrolled in a study where the individual received CTNS-RD-04 will be offered participation in the CTNS-RD-04-LTF01 study. The Baseline visit for the CTNS-RD-04-LTF01 study will likely coincide with the final visit in the parent study. Participants confirmed eligible for the CTNS-RD-04-LTF01 study will be asked to return for study visits at approximately 6-month intervals for the first 4 years and annually thereafter for up to 11 years until a total of 15 years have elapsed during which time continued safety, engraftment, and efficacy of CTNS-RD-04 treatment will be assessed.

ELIGIBILITY:
Inclusion Criteria:

• Participant must have received CTNS-RD-04 in a preceding study

Exclusion Criteria:

• Participant is currently enrolled in an CTNS-RD-04 treatment study. Participants who have either completed, withdrawn, or prematurely discontinued participation for any reason at any time after receiving CTNS-RD-04 are eligible for CTNS RD 04 LTF01 study participation.

Ages: 14 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Participants who received CTNS-RD-04 and agree to comply with the study visit schedule and procedures.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2022-11-14 (Actual); Primary Completion 2036-11-30 (Estimated); Study Completion 2036-11-30 (Estimated)

PRIMARY OUTCOMES:
Incidence of clinically significant Adverse Events (AEs) and Serious Adverse Events (SAEs) | Baseline to Year 15 post gene therapy
Number of participants with clinically relevant abnormalities, as assessed by vital sign (heart rate, pulse rate, and temperature) | Baseline to Year 15 post gene therapy
Number of participants with clinically relevant abnormalities, as assessed by clinical laboratory tests (chemistry and hematology) | Baseline to Year 15 post gene therapy
Number of participants with clinically relevant abnormalities, as assessed by by electrocardiograms (ECGs) (rate, rhythm, intervals) | Baseline to Year 15 post gene therapy

SECONDARY OUTCOMES:
Change from baseline in Corneal cystine crystal score (CCCS) as assessed by in vivo confocal microscopy (IVCM) | Baseline to Year 15 post gene therapy
Change from baseline in Renal glomerular and tubular functions measured by glomerular filtration rate (GFR) | Baseline to Year 15 post gene therapy
Change from baseline in vision function as assessed by ophthalmology exams | Baseline to Year 15 post gene therapy
Change from baseline in grip strength measured by dynamometry | Baseline to Year 15 post gene therapy
Change from baseline in respiratory function measured by spirometry | Baseline to Year 15 post gene therapy
Change from baseline in bone density assessed by dual-energy X-ray absorptiometry (DEXA) | Baseline to Year 15 post gene therapy
Change from baseline in muscle mass assessed by dual-energy X-ray absorptiometry (DEXA) | Baseline to Year 15 post gene therapy
Change from baseline in Endocrine function measured by fasting glucose, thyroid function, and gonadotropin levels | Baseline to Year 15 post gene therapy
Change from baseline in neurological function assessed by neurological exam (mental status, coordination, sensory, reflexes, and visual motor integration) | Baseline to Year 15 post gene therapy
Change from baseline in psychometric function assessed by neurological exam (memory, oromotor function, intelligence quotient (IQ)) | Baseline to Year 15 post gene therapy
Change from baseline in pill/injection count related to cystinosis treatment | Baseline to Year 15 post gene therapy
Change from baseline in Cystinosin (CTNS) as assessed by quantitative Polymerase Chain Reaction (qPCR) | Baseline to Year 15 post gene therapy
Change from baseline in mean Vector Copy Number (VCN) as assessed by quantitative Polymerase Chain Reaction (qPCR) | Baseline to Year 15 post gene therapy
Change from baseline in Cystine levels in leukocytes measured by mass spectrometry | Baseline to Year 15 post gene therapy
Change from baseline in ovarian reserve and menstrual cycle as assessed by anti-Müllerian hormone (AMH) and gynecology exams | Baseline to Year 15 post gene therapy
Change in male reproductive potential as assessed by urology exams (sperm count, motility, and morphology) | Baseline to Year 15 post gene therapy
Absence of Replication Competent Lentivirus (RCL) as assessed by Elisa assay | Baseline to Year 15 post gene therapy

CONTACTS AND LOCATIONS:
Overall Officials: Stephanie Cherqui, PhD, Principal Investigator — University of California, San Diego
Locations (1):
- University of California San Diego, La Jolla, California, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Harrison F, Yeagy BA, Rocca CJ, Kohn DB, Salomon DR, Cherqui S. Hematopoietic stem cell gene therapy for the multisystemic lysosomal storage disorder cystinosis. Mol Ther. 2013 Feb;21(2):433-44. doi: 10.1038/mt.2012.214. Epub 2012 Oct 23. PMID 23089735
- [Result] Naphade S, Sharma J, Gaide Chevronnay HP, Shook MA, Yeagy BA, Rocca CJ, Ur SN, Lau AJ, Courtoy PJ, Cherqui S. Brief reports: Lysosomal cross-correction by hematopoietic stem cell-derived macrophages via tunneling nanotubes. Stem Cells. 2015 Jan;33(1):301-9. doi: 10.1002/stem.1835. PMID 25186209